CLINICAL TRIAL: NCT02516423
Title: Solitary Plasmacytoma of Bone: Randomized Phase III Trial to Evaluate Treatment With Adjuvant Systemic Treatment and Zoledronic Acid Versus Zoledronic Acid After Definite Radiation Therapy
Brief Title: Ixazomib Citrate, Lenalidomide, Dexamethasone, and Zoledronic Acid or Zoledronic Acid Alone After Radiation Therapy in Treating Patients With Solitary Plasmacytoma of Bone
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Alliance for Clinical Trials in Oncology (Other)
Collaborators: National Cancer Institute (NCI) (NIH); Millennium Pharmaceuticals, Inc. (Industry); Biologics, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: A061402; NCI-2015-00323 (Registry Identifier: NCI Clinical Trials Reporting Program); U10CA180821 (NIH)
Record Dates: First submitted 2015-08-04; First posted 2015-08-05 (Estimated); Last update posted 2021-08-17 (Actual); Status verified 2021-08

CONDITIONS: Solitary Osseous Plasmacytoma
MeSH Terms: interventions — ixazomib; Lenalidomide; Dexamethasone; Zoledronic Acid

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- ixazomib + lenalidomide + dexamethasone + zoledronic acid (Experimental): Patients receive 4 mg ixazomib by mouth on days 1, 8 and 15. Patients also receive 15 mg lenalidomide by mouth on days 1-21, 12 mg dexamethasone by mouth on days 1, 8, 15, and 22 and zoledronic acid (dose based on creatinine clearance on day 1) IV infusion on day 1. Patients receive treatment every 28 days for a maximum of 6 cycles.
  Interventions: Drug: ixazomib; Drug: lenalidomide; Drug: dexamethasone; Drug: zoledronic acid
- zoledronic acid (Active Comparator): Patients receive zoledronic acid (dose based on creatinine clearance on day 1) IV on day 1. Patients receive treatment every 28 days for a maximum of 6 cycles.
  Interventions: Drug: zoledronic acid

INTERVENTIONS:
Drug: ixazomib — oral
  Arms: ixazomib + lenalidomide + dexamethasone + zoledronic acid
Drug: lenalidomide — oral
  Arms: ixazomib + lenalidomide + dexamethasone + zoledronic acid
Drug: dexamethasone — oral
  Arms: ixazomib + lenalidomide + dexamethasone + zoledronic acid
Drug: zoledronic acid — IV

SUMMARY:
This randomized phase III trial compares ixazomib citrate, lenalidomide, dexamethasone and zoledronic acid with zoledronic acid alone to see how well they work when given after radiation therapy in treating patients with solitary plasmacytoma of bone. Ixazomib citrate may stop the growth of cancer cells by blocking some of the enzymes needed for cell growth. Lenalidomide may help the immune system kill abnormal blood cells or cancer cells. Dexamethasone is a drug used in chemotherapy that may cause tumor cells to die. Zoledronic acid may prevent bone fractures and reduce bone pain, and may also improve survival. Standard treatment for this cancer is radiation therapy alone. It is not yet known whether ixazomib citrate, lenalidomide, dexamethasone and zoledronic acid or zoledronic acid alone is more effective, and whether adding these treatments after radiation therapy is more effective than radiation therapy alone in treating patients with solitary plasmacytoma of bone.

DETAILED DESCRIPTION:
This phase III randomized clinical trial was designed to assess the impact of the addition of ixazomib, lenalidomide, and dexamethasone to zoledronic acid the multiple myeloma progression rate at 5 years. A dynamic allocation procedure will be used to allocate an equal number of patients to each of the treatment arms. This procedure will balance the number of patients which falls into each of the following categories between the two treatment arms:

1. % of abnormal plasma cells in the bone marrow: 5-9%
2. age < 60; % of abnormal plasma cells in the bone marrow < 5%; and monoclonal protein/clonal light chains present in the blood or urine
3. age < 60; % of abnormal plasma cells in the bone marrow < 5% and no monoclonal protein/clonal light chains present in the blood or urine, (MRD+) minimal residual disease
4. age ≥ 60; % of abnormal plasma cells in the bone marrow < 5%; and monoclonal protein/clonal light chains present in the blood or urine
5. age ≥ 60; % of abnormal plasma cells in the bone marrow < 5% and no monoclonal protein/clonal light chains present in the blood or urine, (MRD+) minimal residual disease

The primary and secondary objectives are described below.

Primary objective

To assess whether ixazomib, lenalidomide, dexamethasone with zoledronic acid is more promising than zoledronic acid alone in increasing the time before progression to multiple myeloma.

Secondary objectives

1. To assess changes in minimal residual disease [MRD] by flow cytometry from study entry, at the completion of treatment, and at 1 year post registration.
2. To assess whether ixazomib, lenalidomide, dexamethasone with zoledronic acid is more promising than zoledronic acid alone in extending overall survival.
3. To examine the pharmacodynamics effects of treatment on biochemical markers of bone formation (osteocalcin bone-specific alkaline phosphatase), resorption (serum CTX), and metabolism (OPG).

Follow-up requirements after documentation of progression to multiple myeloma includes a maximum of five years following registration.

ELIGIBILITY:
Pre-registration eligibility criteria (Step 0)

1. Documentation of Disease: Histologic Documentation of Solitary Bone Plasmacytoma

   1. For patients pre-registering after the completion of radiation therapy, documentation of a bone marrow aspirate and biopsy containing <10% clonal plasma cells done at most 28 days prior to start of radiation therapy
   2. For patients pre-registering before the start of radiation therapy, radiation therapy scheduled to begin at most 28 days after a bone marrow aspirate and biopsy were performed containing <10% clonal plasma cells
   3. Participants must have disease that is measurable by either serum or urine evaluation of the monoclonal component or by assay of serum free light chains or by minimal residual detection. Measurable disease is defined as one or more of the following:

      * serum M protein > 0.5 G/DL, or
      * urine M protein >200 MG/24H, and/or
      * serum FLC assay: involved FLC level > 10 MG/DL with abnormal serum FLC ratio
      * ≥ 50 Plasma cells detectable by multicolor flow cytometry, at a sensitive level of 10^-4
2. Age ≥ 18 years
3. ECOG Performance Status 0-2

Registration Eligibility Criteria (Step 1)

1. Documentation of Disease:

   1. No lytic lesions on skeletal survey and whole body PET/CT other than a single lesion associated with solitary bone plasmacytoma within 28 days prior to registration.
   2. Participants must have disease that is measurable by either serum or urine evaluation of the monoclonal component or by assay of serum free light chains or by minimal residual detection. Measurable disease is defined as one or more of the following:

      * serum M protein > 0.5 G/DL, or
      * urine M protein >200 MG/24H, and/or
      * serum FLC assay: involved FLC level > 10 MG/DL with abnormal serum FLC ratio
      * ≥ 50 Plasma cells detectable by multicolor flow cytometry, at a sensitive level of 10^-4
2. Prior Treatment

   1. No major surgery within 21 days of registration with stabilization or resolution of surgical adverse events.
   2. No investigational agent within 21 days prior to registration
   3. No ongoing therapy with corticosteroids greater than 10 mg of prednisone or its equivalent per day. Please note: Inhaled and topical steroids are permitted.
   4. No prior proteasome inhibitor or IMiD use.
   5. Prior bisphosphonate use is permitted.
   6. For all patients:

      * Radiation dose should range from 4500 cGy to 6000 cGy
      * No treatment for this disease following radiation therapy
      * Registration must be completed within 90 days of completion of radiation therapy.
3. Not pregnant and not nursing, because this study involves an investigational agent whose genotoxic, mutagenic and teratogenic effects on the developing fetus and newborn are unknown and an agent that has known genotoxic, mutagenic and teratogenic effects.

   1. Females of childbearing potential (FCBP), defined as a sexually mature female who 1) has not undergone a hysterectomy or bilateral oophorectomy or 2) has not been naturally postmenopausal for at least 24 consecutive months that is, has not had menses at any time in the preceding 24 consecutive months:

      * must have a negative serum or urine pregnancy test with a sensitivity of at least 50 mIU/mL within 10 - 14 days prior to and again within 24 hours of starting lenalidomide.
      * must either commit to continued abstinence from heterosexual intercourse or begin TWO acceptable methods of birth control, one highly effective method and one additional effective method AT THE SAME TIME, at least 28 days before she starts taking lenalidomide.
      * must agree to ongoing pregnancy testing.
   2. Men must agree to use a latex condom during sexual contact with a FCBP even if they have had a vasectomy.
4. ECOG Performance Status 0-2
5. Required Initial Laboratory Values within 14 days of registration:

   1. Absolute Neutrophil Count (ANC) ≥ 1,500/mm^3
   2. Platelet Count ≥ 75,000/mm^3
   3. Hemoglobin ≥ 10 g/dL
   4. Serum Creatinine < 2.0 mg/dL [176.8 µmol/liter]
   5. Serum calcium ≤ 11.5 mg/dL
   6. Calc. Creatinine Clearance > 50 mL/min
   7. Bilirubin ≤ 1.5 x upper limits of normal (ULN)
   8. AST ≤ 2.5 x upper limits of normal (ULN)
6. Intercurrent or Recent Illness

   1. If history of prior malignancy, subject should be in complete remission for ≥ 5 years at the time of registration (with the exception of basal cell or squamous cell carcinoma of the skin treated with local resection).
   2. HIV + patients are eligible provided they meet the other eligibility criteria and:

      * CD4+ cells are ≥ 250/mm^3
      * There is no history of AIDS defining conditions other than historically low CD4+ cell count.
      * The following antiretroviral agents are not allowed: zidovudine, stavudine, protease inhibitors, combination pills with pharmacologic boosters.
      * Recommended antiretroviral regimens to avoid PK interactions include strand integrase inhibitors with nucleoside and non-nucleoside reverse transcriptase inhibitors (for example, dolutegravir given with tenofovir and emtricitabine).
   3. Patients with HBV infection are eligible provided they meet the other eligibility criteria and:

      * There is no evidence of hepatic damage related to HBV infection.
      * They have had consistently suppressed HBV viral load to undetectable levels by PCR for a minimum of 12 months.
   4. Patients with HCV infection are eligible provided they meet the other eligibility criteria and:

      * They have previously undergone curative therapy and have no evidence of active HCV infection.
      * They have no evidence of liver damage owing to prior HCV infection.

      Patients with active HCV infection should be referred for HCV treatment and standard radiotherapy for the plasmacytoma.
   5. Patients cannot have:

      * Known allergy to boron or excipients in the formulation.
      * Known GI disease or GI procedure that could interfere with the oral absorption or tolerance of study drugs including difficulty swallowing.
      * Infection requiring systemic antibiotic therapy or other serious infection within 14 days before registration.
      * Diarrhea ≥ Grade 1, based on the NCI CTCAE categorization within 14 days of registration
      * Life-threatening illness unrelated to cancer
      * The development of erythema nodosum if characterized by a desquamating rash while taking thalidomide, pomalidomide, or similar drugs.
7. Peripheral Neuropathy: ≤ Grade 2 Peripheral Neuropathy
8. Adequate cardiac function, defined as:

   1. No cardiac arrhythmias within 182 days of registration.
   2. No congestive heart failure (CHF) within 182 days of registration.
   3. No angina or myocardial infarction within 182 days of registration. In view of potential cardiac risk with lenalidomide, patients with stable angina will be excluded.
9. Concomitant Treatment: Patients cannot be on systemic treatment with strong inhibitors of CYP1A2 (fluvoxamine, enoxacin), strong inhibitors of CYP3A (clarithromycin, telithromycin, itraconazole, voriconazole, ketoconazole, nefazodone) or strong CYP3A inducers (rifampin, rifapentine, rifabutin, carbamazepine, phenytoin, phenobarbital) within 14 days of registration.
10. QT c< 470 milliseconds (msec) on a 12-lead ECG ≤ 28 days before registration
11. Dental evaluation within 35 days of registration: Complete dental exam; complete elimination of dental and periodontal pathology including crowns on teeth susceptible to fracture, extraction of non-restorable or periodontally uncorrectable teeth; creation of an oral environment that the patient can efficiently maintain in a high state of health; and oral hygiene instruction to maintain excellent oral health.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 11 (Actual)
Dates: Start 2015-12 (Actual); Primary Completion 2024-09 (Estimated)

PRIMARY OUTCOMES:
Progression-free survival rate | at 5 years

SECONDARY OUTCOMES:
Changes in minimal residual disease from study entry to the completion of adjuvant treatment (approximately six months post-registration) and at 1 year post-registration | at 6 and 12 months post-registration
Clinical response rate at 12 months post-registration using whole body PET/CT | at 12 months post-registration

CONTACTS AND LOCATIONS:
Overall Officials: Anuj Mahindra, MD, Study Chair — Scripps Health
Locations (388):
- United States (388):
  - Anchorage Associates in Radiation Medicine, Anchorage, Alaska
  - Anchorage Radiation Therapy Center, Anchorage, Alaska
  - Alaska Breast Care and Surgery LLC, Anchorage, Alaska
  - Alaska Oncology and Hematology LLC, Anchorage, Alaska
  - Alaska Women's Cancer Care, Anchorage, Alaska
  - Anchorage Oncology Centre, Anchorage, Alaska
  - Katmai Oncology Group, Anchorage, Alaska
  - Providence Alaska Medical Center, Anchorage, Alaska
  - Providence Saint Joseph Medical Center/Disney Family Cancer Center, Burbank, California
  - University Oncology Associates, Clovis, California
  - Epic Care-Dublin, Dublin, California
  - Bay Area Breast Surgeons Inc, Emeryville, California
  - Epic Care Partners in Cancer Care, Emeryville, California
  - California Cancer Center - Fresno, Fresno, California
  - Scripps Cancer Center, La Jolla, California
  - Contra Costa Regional Medical Center, Martinez, California
  - Alta Bates Summit Medical Center - Summit Campus, Oakland, California
  - Bay Area Tumor Institute, Oakland, California
  - Epic Care Cyberknife Center, Walnut Creek, California
  - Grand Valley Oncology, Grand Junction, Colorado
  - Saint Alphonsus Cancer Care Center-Boise, Boise, Idaho
  - Saint Luke's Mountain States Tumor Institute, Boise, Idaho
  - Saint Alphonsus Cancer Care Center-Caldwell, Caldwell, Idaho
  - Kootenai Medical Center, Coeur d'Alene, Idaho
  - Walter Knox Memorial Hospital, Emmett, Idaho
  - Saint Luke's Mountain States Tumor Institute - Fruitland, Fruitland, Idaho
  - Idaho Urologic Institute-Meridian, Meridian, Idaho
  - Saint Luke's Mountain States Tumor Institute - Meridian, Meridian, Idaho
  - Saint Alphonsus Medical Center-Nampa, Nampa, Idaho
  - Saint Luke's Mountain States Tumor Institute - Nampa, Nampa, Idaho
  - Kootenai Cancer Center, Post Falls, Idaho
  - Kootenai Cancer Clinic, Sandpoint, Idaho
  - Saint Luke's Mountain States Tumor Institute-Twin Falls, Twin Falls, Idaho
  - Rush - Copley Medical Center, Aurora, Illinois
  - Saint Joseph Medical Center, Bloomington, Illinois
  - Illinois CancerCare-Bloomington, Bloomington, Illinois
  - Illinois CancerCare-Canton, Canton, Illinois
  - Memorial Hospital of Carbondale, Carbondale, Illinois
  - SIH Cancer Institute, Carterville, Illinois
  - Illinois CancerCare-Carthage, Carthage, Illinois
  - Centralia Oncology Clinic, Centralia, Illinois
  - Rush University Medical Center, Chicago, Illinois
  - Carle on Vermilion, Danville, Illinois
  - Cancer Care Specialists of Illinois - Decatur, Decatur, Illinois
  - Decatur Memorial Hospital, Decatur, Illinois
  - Carle Physician Group-Effingham, Effingham, Illinois
  - Crossroads Cancer Center, Effingham, Illinois
  - Illinois CancerCare-Eureka, Eureka, Illinois
  - Illinois CancerCare-Galesburg, Galesburg, Illinois
  - Western Illinois Cancer Treatment Center, Galesburg, Illinois
  - Illinois CancerCare-Kewanee Clinic, Kewanee, Illinois
  - Illinois CancerCare-Macomb, Macomb, Illinois
  - Carle Physician Group-Mattoon/Charleston, Mattoon, Illinois
  - Good Samaritan Regional Health Center, Mount Vernon, Illinois
  - Illinois CancerCare-Ottawa Clinic, Ottawa, Illinois
  - Radiation Oncology of Northern Illinois, Ottawa, Illinois
  - Illinois CancerCare-Pekin, Pekin, Illinois
  - OSF Saint Francis Radiation Oncology at Pekin Cancer Treatment Center, Pekin, Illinois
  - Illinois CancerCare-Peoria, Peoria, Illinois
  - OSF Saint Francis Radiation Oncology at Peoria Cancer Center, Peoria, Illinois
  - Methodist Medical Center of Illinois, Peoria, Illinois
  - OSF Saint Francis Medical Center, Peoria, Illinois
  - Illinois CancerCare-Peru, Peru, Illinois
  - Valley Radiation Oncology, Peru, Illinois
  - Illinois CancerCare-Princeton, Princeton, Illinois
  - Central Illinois Hematology Oncology Center, Springfield, Illinois
  - Southern Illinois University School of Medicine, Springfield, Illinois
  - Springfield Clinic, Springfield, Illinois
  - Memorial Medical Center, Springfield, Illinois
  - Cancer Care Specialists of Illinois-Swansea, Swansea, Illinois
  - Southwest Illinois Health Services LLP, Swansea, Illinois
  - Carle Cancer Center, Urbana, Illinois
  - The Carle Foundation Hospital, Urbana, Illinois
  - Rush-Copley Healthcare Center, Yorkville, Illinois
  - Deaconess Clinic Downtown, Evansville, Indiana
  - Parkview Hospital Randallia, Fort Wayne, Indiana
  - Indiana University/Melvin and Bren Simon Cancer Center, Indianapolis, Indiana
  - Springmill Medical Center, Indianapolis, Indiana
  - Franciscan Saint Anthony Health-Michigan City, Michigan City, Indiana
  - Woodland Cancer Care Center, Michigan City, Indiana
  - Memorial Regional Cancer Center Day Road, Mishawaka, Indiana
  - Chancellor Center for Oncology, Newburgh, Indiana
  - Reid Health, Richmond, Indiana
  - Memorial Hospital of South Bend, South Bend, Indiana
  - Cancer Center of Kansas - Chanute, Chanute, Kansas
  - Cancer Center of Kansas - Dodge City, Dodge City, Kansas
  - Cancer Center of Kansas - El Dorado, El Dorado, Kansas
  - Cancer Center of Kansas - Fort Scott, Fort Scott, Kansas
  - Cancer Center of Kansas-Independence, Independence, Kansas
  - Cancer Center of Kansas-Kingman, Kingman, Kansas
  - Lawrence Memorial Hospital, Lawrence, Kansas
  - Cancer Center of Kansas-Liberal, Liberal, Kansas
  - Cancer Center of Kansas-Manhattan, Manhattan, Kansas
  - Cancer Center of Kansas - McPherson, McPherson, Kansas
  - Cancer Center of Kansas - Newton, Newton, Kansas
  - Cancer Center of Kansas - Parsons, Parsons, Kansas
  - Cancer Center of Kansas - Pratt, Pratt, Kansas
  - Cancer Center of Kansas - Salina, Salina, Kansas
  - Cancer Center of Kansas - Wellington, Wellington, Kansas
  - Associates In Womens Health, Wichita, Kansas
  - Cancer Center of Kansas-Wichita Medical Arts Tower, Wichita, Kansas
  - Cancer Center of Kansas - Wichita, Wichita, Kansas
  - Wesley Medical Center, Wichita, Kansas
  - Cancer Center of Kansas - Winfield, Winfield, Kansas
  - Oncology Hematology Care Inc-Crestview, Crestview Hills, Kentucky
  - Ochsner Medical Center Jefferson, New Orleans, Louisiana
  - Harold Alfond Center for Cancer Care, Augusta, Maine
  - Eastern Maine Medical Center, Bangor, Maine
  - Lafayette Family Cancer Center-EMMC, Brewer, Maine
  - Massachusetts General Hospital Cancer Center, Boston, Massachusetts
  - Dana-Farber Cancer Institute, Boston, Massachusetts
  - Mercy Medical Center, Springfield, Massachusetts
  - Hickman Cancer Center, Adrian, Michigan
  - Saint Joseph Mercy Hospital, Ann Arbor, Michigan
  - Bronson Battle Creek, Battle Creek, Michigan
  - IHA Hematology Oncology Consultants-Brighton, Brighton, Michigan
  - Saint Joseph Mercy Brighton, Brighton, Michigan
  - Henry Ford Cancer Institute?Downriver, Brownstown, Michigan
  - IHA Hematology Oncology Consultants-Canton, Canton, Michigan
  - Saint Joseph Mercy Canton, Canton, Michigan
  - Caro Cancer Center, Caro, Michigan
  - IHA Hematology Oncology Consultants-Chelsea, Chelsea, Michigan
  - Saint Joseph Mercy Chelsea, Chelsea, Michigan
  - Hematology Oncology Consultants-Clarkston, Clarkston, Michigan
  - Newland Medical Associates-Clarkston, Clarkston, Michigan
  - Henry Ford Macomb Hospital-Clinton Township, Clinton Township, Michigan
  - Beaumont Hospital-Dearborn, Dearborn, Michigan
  - Henry Ford Medical Center-Fairlane, Dearborn, Michigan
  - Henry Ford Hospital, Detroit, Michigan
  - Ascension Saint John Hospital, Detroit, Michigan
  - Great Lakes Cancer Management Specialists-Doctors Park, East China Township, Michigan
  - Genesee Cancer and Blood Disease Treatment Center, Flint, Michigan
  - Genesee Hematology Oncology PC, Flint, Michigan
  - Genesys Hurley Cancer Institute, Flint, Michigan
  - Hurley Medical Center, Flint, Michigan
  - Mercy Health Saint Mary's, Grand Rapids, Michigan
  - Spectrum Health at Butterworth Campus, Grand Rapids, Michigan
  - Great Lakes Cancer Management Specialists-Van Elslander Cancer Center, Grosse Pointe Woods, Michigan
  - Lymphoma Clinic of Michigan, Grosse Pointe Woods, Michigan
  - Michigan Breast Specialists-Grosse Pointe Woods, Grosse Pointe Woods, Michigan
  - Allegiance Health, Jackson, Michigan
  - Bronson Methodist Hospital, Kalamazoo, Michigan
  - West Michigan Cancer Center, Kalamazoo, Michigan
  - Borgess Medical Center, Kalamazoo, Michigan
  - Sparrow Hospital, Lansing, Michigan
  - Hope Cancer Clinic, Livonia, Michigan
  - Saint Mary Mercy Hospital, Livonia, Michigan
  - Great Lakes Cancer Management Specialists-Macomb Medical Campus, Macomb, Michigan
  - Michigan Breast Specialists-Macomb Township, Macomb, Michigan
  - Saint Mary's Oncology/Hematology Associates of Marlette, Marlette, Michigan
  - Toledo Clinic Cancer Centers-Monroe, Monroe, Michigan
  - Mercy Health Mercy Campus, Muskegon, Michigan
  - Lakeland Hospital Niles, Niles, Michigan
  - Ascension Providence Hospitals - Novi, Novi, Michigan
  - Henry Ford Medical Center-Columbus, Novi, Michigan
  - 21st Century Oncology-Pontiac, Pontiac, Michigan
  - Hope Cancer Center, Pontiac, Michigan
  - Newland Medical Associates-Pontiac, Pontiac, Michigan
  - Saint Joseph Mercy Oakland, Pontiac, Michigan
  - Spectrum Health Reed City Hospital, Reed City, Michigan
  - Great Lakes Cancer Management Specialists-Rochester Hills, Rochester Hills, Michigan
  - Saint Mary's of Michigan, Saginaw, Michigan
  - Oncology Hematology Associates of Saginaw Valley PC, Saginaw, Michigan
  - Lakeland Medical Center Saint Joseph, Saint Joseph, Michigan
  - Marie Yeager Cancer Center, Saint Joseph, Michigan
  - Ascension Providence Hospitals - Southfield, Southfield, Michigan
  - Bhadresh Nayak MD PC-Sterling Heights, Sterling Heights, Michigan
  - Saint Joseph Health System-Tawas City, Tawas City, Michigan
  - Munson Medical Center, Traverse City, Michigan
  - Advanced Breast Care Center PLLC, Warren, Michigan
  - Bhadresh Nayak MD PC-Warren, Warren, Michigan
  - Great Lakes Cancer Management Specialists-Macomb Professional Building, Warren, Michigan
  - Macomb Hematology Oncology PC, Warren, Michigan
  - Michigan Breast Specialists-Warren, Warren, Michigan
  - Saint John Macomb-Oakland Hospital, Warren, Michigan
  - Henry Ford West Bloomfield Hospital, West Bloomfield, Michigan
  - Saint Mary's Oncology/Hematology Associates of West Branch, West Branch, Michigan
  - Metro Health Hospital, Wyoming, Michigan
  - Huron Gastroenterology PC, Ypsilanti, Michigan
  - IHA Hematology Oncology Consultants-Ann Arbor, Ypsilanti, Michigan
  - Sanford Joe Lueken Cancer Center, Bemidji, Minnesota
  - Essentia Health Saint Joseph's Medical Center, Brainerd, Minnesota
  - Essentia Health - Deer River Clinic, Deer River, Minnesota
  - Essentia Health Saint Mary's - Detroit Lakes Clinic, Detroit Lakes, Minnesota
  - Essentia Health Cancer Center, Duluth, Minnesota
  - Essentia Health Saint Mary's Medical Center, Duluth, Minnesota
  - Miller-Dwan Hospital, Duluth, Minnesota
  - Lake Region Healthcare Corporation-Cancer Care, Fergus Falls, Minnesota
  - Essentia Health - Fosston, Fosston, Minnesota
  - Essentia Health Hibbing Clinic, Hibbing, Minnesota
  - Essentia Health - Park Rapids, Park Rapids, Minnesota
  - Mayo Clinic, Rochester, Minnesota
  - Essentia Health Sandstone, Sandstone, Minnesota
  - Sanford Thief River Falls Medical Center, Thief River Falls, Minnesota
  - Essentia Health Virginia Clinic, Virginia, Minnesota
  - Sanford Cancer Center Worthington, Worthington, Minnesota
  - University of Mississippi Medical Center, Jackson, Mississippi
  - Saint Louis Cancer and Breast Institute-Ballwin, Ballwin, Missouri
  - Central Care Cancer Center - Bolivar, Bolivar, Missouri
  - Parkland Health Center-Bonne Terre, Bonne Terre, Missouri
  - Cox Cancer Center Branson, Branson, Missouri
  - Saint Francis Medical Center, Cape Girardeau, Missouri
  - Southeast Cancer Center, Cape Girardeau, Missouri
  - Capital Region Southwest Campus, Jefferson City, Missouri
  - Freeman Health System, Joplin, Missouri
  - Mercy Hospital Joplin, Joplin, Missouri
  - Delbert Day Cancer Institute at PCRMC, Rolla, Missouri
  - Mercy Clinic-Rolla-Cancer and Hematology, Rolla, Missouri
  - Heartland Regional Medical Center, Saint Joseph, Missouri
  - Sainte Genevieve County Memorial Hospital, Sainte Genevieve, Missouri
  - Mercy Hospital Springfield, Springfield, Missouri
  - CoxHealth South Hospital, Springfield, Missouri
  - Saint Louis Cancer and Breast Institute-South City, St Louis, Missouri
  - Missouri Baptist Medical Center, St Louis, Missouri
  - Mercy Hospital Saint Louis, St Louis, Missouri
  - Missouri Baptist Sullivan Hospital, Sullivan, Missouri
  - Missouri Baptist Outpatient Center-Sunset Hills, Sunset Hills, Missouri
  - Mercy Hospital Washington, Washington, Missouri
  - Community Hospital of Anaconda, Anaconda, Montana
  - Billings Clinic Cancer Center, Billings, Montana
  - Saint Vincent Healthcare, Billings, Montana
  - Bozeman Deaconess Hospital, Bozeman, Montana
  - Saint James Community Hospital and Cancer Treatment Center, Butte, Montana
  - Benefis Healthcare- Sletten Cancer Institute, Great Falls, Montana
  - Great Falls Clinic, Great Falls, Montana
  - Saint Peter's Community Hospital, Helena, Montana
  - Kalispell Regional Medical Center, Kalispell, Montana
  - Saint Patrick Hospital - Community Hospital, Missoula, Montana
  - Community Medical Hospital, Missoula, Montana
  - Dartmouth Hitchcock Medical Center, Lebanon, New Hampshire
  - Norris Cotton Cancer Center-Nashua, Nashua, New Hampshire
  - Roswell Park Cancer Institute, Buffalo, New York
  - Wake Forest University Health Sciences, Winston-Salem, North Carolina
  - Sanford Bismarck Medical Center, Bismarck, North Dakota
  - Essentia Health Cancer Center-South University Clinic, Fargo, North Dakota
  - Sanford South University Medical Center, Fargo, North Dakota
  - Roger Maris Cancer Center, Fargo, North Dakota
  - Sanford Broadway Medical Center, Fargo, North Dakota
  - Essentia Health - Jamestown Clinic, Jamestown, North Dakota
  - Indu and Raj Soin Medical Center, Beavercreek, Ohio
  - Strecker Cancer Center-Belpre, Belpre, Ohio
  - Dayton Physicians LLC-Miami Valley South, Centerville, Ohio
  - Miami Valley Hospital South, Centerville, Ohio
  - Adena Regional Medical Center, Chillicothe, Ohio
  - Oncology Hematology Care Inc-Eden Park, Cincinnati, Ohio
  - Oncology Hematology Care Inc-Mercy West, Cincinnati, Ohio
  - Oncology Hematology Care Inc - Anderson, Cincinnati, Ohio
  - Oncology Hematology Care Inc-Kenwood, Cincinnati, Ohio
  - Oncology Hematology Care Inc-Blue Ash, Cincinnati, Ohio
  - Mount Carmel East Hospital, Columbus, Ohio
  - Columbus Oncology and Hematology Associates Inc, Columbus, Ohio
  - Riverside Methodist Hospital, Columbus, Ohio
  - Grant Medical Center, Columbus, Ohio
  - The Mark H Zangmeister Center, Columbus, Ohio
  - Mount Carmel Health Center West, Columbus, Ohio
  - Doctors Hospital, Columbus, Ohio
  - Good Samaritan Hospital - Dayton, Dayton, Ohio
  - Miami Valley Hospital, Dayton, Ohio
  - Dayton Physicians LLC-Samaritan North, Dayton, Ohio
  - Miami Valley Hospital North, Dayton, Ohio
  - Delaware Health Center-Grady Cancer Center, Delaware, Ohio
  - Delaware Radiation Oncology, Delaware, Ohio
  - Grady Memorial Hospital, Delaware, Ohio
  - Oncology Hematology Care Inc-Healthplex, Fairfield, Ohio
  - Armes Family Cancer Center, Findlay, Ohio
  - Blanchard Valley Hospital, Findlay, Ohio
  - Orion Cancer Care, Findlay, Ohio
  - Atrium Medical Center-Middletown Regional Hospital, Franklin, Ohio
  - Dayton Physicians LLC-Atrium, Franklin, Ohio
  - Dayton Physicians LLC-Wayne, Greenville, Ohio
  - Wayne Hospital, Greenville, Ohio
  - Greater Dayton Cancer Center, Kettering, Ohio
  - First Dayton Cancer Care, Kettering, Ohio
  - Kettering Medical Center, Kettering, Ohio
  - Fairfield Medical Center, Lancaster, Ohio
  - OhioHealth Mansfield Hospital, Mansfield, Ohio
  - Marietta Memorial Hospital, Marietta, Ohio
  - OhioHealth Marion General Hospital, Marion, Ohio
  - Toledo Clinic Cancer Centers-Maumee, Maumee, Ohio
  - Toledo Radiation Oncology at Northwest Ohio Onocolgy Center, Maumee, Ohio
  - Dayton Physicians LLC-Signal Point, Middletown, Ohio
  - Knox Community Hospital, Mount Vernon, Ohio
  - Licking Memorial Hospital, Newark, Ohio
  - Newark Radiation Oncology, Newark, Ohio
  - Saint Charles Hospital, Oregon, Ohio
  - Mercy Health Perrysburg Cancer Center, Perrysburg, Ohio
  - Southern Ohio Medical Center, Portsmouth, Ohio
  - Dayton Physicians LLC-Wilson, Sidney, Ohio
  - Springfield Regional Cancer Center, Springfield, Ohio
  - Springfield Regional Medical Center, Springfield, Ohio
  - Mercy Saint Anne Hospital, Toledo, Ohio
  - Toledo Clinic Cancer Centers-Toledo, Toledo, Ohio
  - Dayton Physicians LLC-Upper Valley, Troy, Ohio
  - Upper Valley Medical Center, Troy, Ohio
  - Saint Ann's Hospital, Westerville, Ohio
  - Genesis Healthcare System Cancer Care Center, Zanesville, Ohio
  - Cancer Centers of Southwest Oklahoma Research, Lawton, Oklahoma
  - University of Oklahoma Health Sciences Center, Oklahoma City, Oklahoma
  - Mercy Hospital Oklahoma City, Oklahoma City, Oklahoma
  - Saint Alphonsus Medical Center-Baker City, Baker City, Oregon
  - Saint Charles Health System, Bend, Oregon
  - Clackamas Radiation Oncology Center, Clackamas, Oregon
  - Providence Oncology and Hematology Care Southeast, Clackamas, Oregon
  - Bay Area Hospital, Coos Bay, Oregon
  - Providence Newberg Medical Center, Newberg, Oregon
  - Saint Alphonsus Medical Center-Ontario, Ontario, Oregon
  - Providence Willamette Falls Medical Center, Oregon City, Oregon
  - Providence Portland Medical Center, Portland, Oregon
  - Providence Saint Vincent Medical Center, Portland, Oregon
  - Saint Charles Health System-Redmond, Redmond, Oregon
  - Lehigh Valley Hospital-Cedar Crest, Allentown, Pennsylvania
  - Lehigh Valley Hospital - Muhlenberg, Bethlehem, Pennsylvania
  - Geisinger Medical Center, Danville, Pennsylvania
  - Geisinger Medical Center-Cancer Center Hazleton, Hazleton, Pennsylvania
  - Geisinger Medical Oncology-Lewisburg, Lewisburg, Pennsylvania
  - Lewistown Hospital, Lewistown, Pennsylvania
  - Geisinger Cancer Services-Pottsville, Pottsville, Pennsylvania
  - Community Medical Center, Scranton, Pennsylvania
  - Geisinger Medical Oncology-Selinsgrove, Selinsgrove, Pennsylvania
  - Geisinger Medical Group, State College, Pennsylvania
  - Geisinger Wyoming Valley/Henry Cancer Center, Wilkes-Barre, Pennsylvania
  - Gibbs Cancer Center-Gaffney, Gaffney, South Carolina
  - Saint Francis Hospital, Greenville, South Carolina
  - Saint Francis Cancer Center, Greenville, South Carolina
  - Gibbs Cancer Center-Pelham, Greer, South Carolina
  - Spartanburg Medical Center, Spartanburg, South Carolina
  - MGC Hematology Oncology-Union, Union, South Carolina
  - Sanford Cancer Center Oncology Clinic, Sioux Falls, South Dakota
  - Sanford USD Medical Center - Sioux Falls, Sioux Falls, South Dakota
  - Parkland Memorial Hospital, Dallas, Texas
  - UT Southwestern/Simmons Cancer Center-Dallas, Dallas, Texas
  - UT Southwestern/Simmons Cancer Center-Fort Worth, Fort Worth, Texas
  - M D Anderson Cancer Center, Houston, Texas
  - Farmington Health Center, Farmington, Utah
  - Huntsman Cancer Institute/University of Utah, Salt Lake City, Utah
  - South Jordan Health Center, South Jordan, Utah
  - Norris Cotton Cancer Center-North, Saint Johnsbury, Vermont
  - Danville Hematology Oncology, Danville, Virginia
  - Danville Regional Medical Center, Danville, Virginia
  - Providence Regional Cancer System-Aberdeen, Aberdeen, Washington
  - Cancer Care Center at Island Hospital, Anacortes, Washington
  - Swedish Cancer Institute-Eastside Oncology Hematology, Bellevue, Washington
  - PeaceHealth Saint Joseph Medical Center, Bellingham, Washington
  - Providence Regional Cancer System-Centralia, Centralia, Washington
  - Swedish Medical Center-Edmonds, Edmonds, Washington
  - Providence Regional Cancer Partnership, Everett, Washington
  - Swedish Cancer Institute-Issaquah, Issaquah, Washington
  - Kadlec Clinic Hematology and Oncology, Kennewick, Washington
  - Providence Regional Cancer System-Lacey, Lacey, Washington
  - PeaceHealth Saint John Medical Center, Longview, Washington
  - Minor and James Medical PLLC, Seattle, Washington
  - Pacific Gynecology Specialists, Seattle, Washington
  - Swedish Medical Center-Ballard Campus, Seattle, Washington
  - Kaiser Permanente Washington, Seattle, Washington
  - Swedish Medical Center-First Hill, Seattle, Washington
  - Swedish Medical Center-Cherry Hill, Seattle, Washington
  - PeaceHealth United General Medical Center, Sedro-Woolley, Washington
  - Providence Regional Cancer System-Shelton, Shelton, Washington
  - Rockwood Cancer Treatment Center-DHEC-Downtown, Spokane, Washington
  - Rockwood North Cancer Treatment Center, Spokane, Washington
  - Rockwood Clinic Cancer Treatment Center-Valley, Spokane Valley, Washington
  - PeaceHealth Southwest Medical Center, Vancouver, Washington
  - Providence Saint Mary Regional Cancer Center, Walla Walla, Washington
  - North Star Lodge Cancer Center at Yakima Valley Memorial Hospital, Yakima, Washington
  - Providence Regional Cancer System-Yelm, Yelm, Washington
  - Ashland Memorial Medical Center, Ashland, Wisconsin
  - Duluth Clinic Ashland, Ashland, Wisconsin
  - Aurora Cancer Care-Southern Lakes VLCC, Burlington, Wisconsin
  - Aurora Health Center-Fond du Lac, Fond du Lac, Wisconsin
  - Aurora Health Care Germantown Health Center, Germantown, Wisconsin
  - Aurora Cancer Care-Grafton, Grafton, Wisconsin
  - Aurora BayCare Medical Center, Green Bay, Wisconsin
  - Aurora Cancer Care-Kenosha South, Kenosha, Wisconsin
  - Gundersen Lutheran Medical Center, La Crosse, Wisconsin
  - Aurora Bay Area Medical Group-Marinette, Marinette, Wisconsin
  - Aurora Cancer Care-Milwaukee, Milwaukee, Wisconsin
  - Aurora Saint Luke's Medical Center, Milwaukee, Wisconsin
  - Aurora Sinai Medical Center, Milwaukee, Wisconsin
  - Vince Lombardi Cancer Clinic - Oshkosh, Oshkosh, Wisconsin
  - Aurora Cancer Care-Racine, Racine, Wisconsin
  - Vince Lombardi Cancer Clinic-Sheboygan, Sheboygan, Wisconsin
  - Aurora Medical Center in Summit, Summit, Wisconsin
  - Vince Lombardi Cancer Clinic-Two Rivers, Two Rivers, Wisconsin
  - Aurora Cancer Care-Milwaukee West, Wauwatosa, Wisconsin
  - Aurora West Allis Medical Center, West Allis, Wisconsin
  - Big Horn Basin Cancer Center, Cody, Wyoming
  - Billings Clinic-Cody, Cody, Wyoming
  - Welch Cancer Center, Sheridan, Wyoming